CLINICAL TRIAL: NCT01359865
Title: The Influence of Anesthetic Technique on Post-operative Pain Scores and Range of Motion in Primary Total Hip Arthroplasty
Brief Title: Comparison of Anesthetic Techniques on Total Hip Arthroplasty
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: change in clinical practice- both surgeons have left the institution
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Jonathan Anson, Assitant professor of Anesthesiology, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: MSHersheyMC
Record Dates: First submitted 2011-05-23; First posted 2011-05-25 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-09

CONDITIONS: Osteoarthritis
Keywords: Total hip arthroplasty; lumbar plexus block; spinal anesthesia; range of motion; Anesthetic Technique; Post-operative Pain Scores
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lumbar plexus Block (No Intervention): This group will recieve pre-operative lumbar plexus block plus general anesthesia
  Interventions: Procedure: Lumbar Plexus Block

INTERVENTIONS:
Procedure: Lumbar Plexus Block — lumbar plexus block followed by a general anesthetic. The lumbar plexus block will be performed by an attending anesthesiologist using ultrasound guidance (for measuring the depth of the psoas compartment) and nerve stimulation. A standardized block solution of 30 mL 0.5% ropivacaine will be injected in fractionated doses when a quadriceps muscle twitch is present to nerve stimulation at <0.50 mA. Fifteen minutes after block completion, the block's effectiveness will be evaluated with an ice test.

SUMMARY:
To compare analgesia and orthopedic rehabilitation milestones in patients receiving either spinal anesthesia (local anesthetic plus opioid) or general endotracheal anesthesia with lumbar plexus block.

DETAILED DESCRIPTION:
To compare analgesia and orthopedic rehabilitation milestones in patients receiving either spinal anesthesia (local anesthetic plus opioid) or general endotracheal anesthesia with lumbar plexus block.

: Total hip arthroplasty (THA) is a common surgery worldwide. Despite the prevalence of this procedure, there is no "gold standard" anesthetic. Several different techniques are utilized. The two most common anesthesia modalities are: 1) spinal anesthesia 2) general anesthesia (with or without a peripheral nerve block). The choice of anesthetic technique is often based on the training and experience of the anesthesia provider, as well as the culture of the institution. Both spinal anesthesia (consisting of local anesthetic and opioid) and general anesthesia (combined with lumbar plexus nerve block) can provide adequate intra-operative anesthesia as well as prolonged post-operative analgesia. The goal of this study is to determine if the choice of one of these two anesthetic techniques influences postoperative pain scores and orthopedic rehabilitation markers in patients undergoing primary THA.

Several studies have compared spinal versus general anesthesia in terms of post-operative pain relief, nausea and vomiting, blood loss, and deep venous thrombosis. Most of these studies did not utilize a lumbar plexus nerve block for postoperative analgesia in the general anesthesia subjects. The investigators are not aware of any randomized, controlled studies examining differences in orthopedic outcomes when THA is performed under spinal anesthesia or general anesthesia with lumbar plexus nerve block. These two anesthetic techniques result in different degrees of intraoperative muscle relaxation which may affect post-operative range of motion. Analgesic differences between the two techniques may also affect range of motion and post-operative ambulation.

The investigators propose to compare post-operative pain scores as a primary outcome in patients receiving either spinal anesthesia (bupivicaine with morphine) or general anesthesia with lumbar plexus block for THA. Orthopedic outcomes, including distance of first ambulation, physical therapy range of motion, and limb length discrepancies will be measured as secondary outcomes. Continuous pulse oximetry and capnograpahy data will be recorded for 24 hours postoperatively on all patients. The incidence of urinary tract infections and post-operative nausea and vomiting between groups will be additional measured outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Elective primary THA
* Surgery by Dr. Fenwick and Dr. Raab
* Anesthesia clinic pre-operative appointment
* ASA I, II, III

Exclusion Criteria:

* Revision THA
* Prior THA on opposite side
* Traumatic hip injury
* Contraindication to neuraxial or regional anesthesia
* History of post-operative nausea and vomiting > 2 prior general anesthetics
* Allergy to local anesthetics, morphine, hydromorphone, dexamethasone, or ondansetron
* History of substance abuse or chronic narcotic use
* Severe degenerative joint disease to non-operative joint impairing ambulation
* Severe back pain or spinal cord stenosis limiting ambulation
* BMI > 40

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-05 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
To compare analgesia and orthopedic rehabilitation milestones (range of motion) in patients receiving either spinal anesthesia (local anesthetic plus opioid) or general endotracheal anesthesia with lumbar plexus block. | Approx one to three month post-op
  On arrival to the adult orthopedic/joint reconstruction ward, a physical therapist will assess the range of motion and document the findings in Powerchart using a pre-existing template. This will be the main primary outcome measure along with ongoing pain scale as part of the orthopedic rehabilitation milestones.

CONTACTS AND LOCATIONS:
Overall Officials: John Anson, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States